CLINICAL TRIAL: NCT00627718
Title: Assessment of Macular Edema Using HRT Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Mila Oh, MD, MUHC
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: BMB 06-029
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; HRT; Macular edema; Screening for disease
MeSH Terms: conditions — Macular Degeneration; Macular Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): All patients with possible neovascular ARMD are assessed with HRT to determined the positive predictive value of the test
  Interventions: Device: HRT screening for macula edema

INTERVENTIONS:
Device: HRT screening for macula edema — HRT screening for macula edema at time of initial diagnosis of macular degeneration

SUMMARY:
Age Related Macular Degeneration (ARMD) is the most common cause of irreversible blindness in people of age 50 or older in the western populations. ARMD has two forms, the wet and the dry forms. The wet form is more serious and can lead to irreversible loss of vision. In the wet form of ARMD, new blood vessels grow under the retina. These blood vessels leak blood and fluid and cause the retina and the macula to swell. So the thickness of the macula increases.

One of the key factors in the treatment of wet ARMD is early diagnosis and treatment to prevent complete visual loss. In this research, we are going to use a technique, called the Heidelberg retinal tomograph (HRT) to measure and compare the thickness of the macula in healthy controls and in patients suspected of having ARMD. HRT is a non-invasive imaging system that uses laser to measure the thickness of the macula. This allows us to come up with a quite simple and easy-to-use technique that helps us to diagnose wet ARMD early and treat it before visual acuity is completely lost.

DETAILED DESCRIPTION:
Introduction: Age-related macular degeneration (ARMD) is a spectrum of related diseases that affects the macula and it has been traditionally classified into early and late stages with its dry (non-exudative) and wet (exudative) forms. Although the advanced form of AMD is less common, the potential visual loss is more significant. The Beaver Dam Eye Study reported that 30% of individuals aged 75 and older have some form of AMD, whereas 7% of those aged 75 and older have an advanced form. Recent studies estimate that 8 million Americans are considered to be at risk for developing advanced ARMD in the next 5 years, whereas 1.75 million are currently affected with the advanced form of the disease.

Wet AMD is characterized by proliferation of abnormal vessels in the choroid. These choroidal neovascular membranes may proliferate into the subretinal space and retina and leak fluid and blood. This fluid may accumulate in the macula area causing macular edema (ME), the final common pathway for visual loss in many diseases. There are currently no treatments that can reverse or repair the destruction and restore visual acuity. The critical time for any intervention is early in the disease, when visual acuity has been minimally affected. Due to the irreversible nature of the disease and a realistic risk of permanent vision loss, there is an increased need to improve the accuracy of identifying the presence and extent of MEvwith a prompt referral to a retina specialist following diagnosis.

ME has traditionally been assessed clinically using a combination of slit lamp biomicroscopy and fluorescein angiography. New imaging techniques such as optical coherence tomography (OCT), the retinal thickness analyser (RTA), and the Heidelberg retinal tomograph (HRT) confocal scanning laser ophthalmoscope facilitate qualitative assessments of the degree of ME. Although OCT has a high sensitivity and specificity for the detection of ME within 500 microns of the fovea, this resolution decreases outside this area. RTA has shown lower sensitivity (57%) for the detection of ME. 4 The Heidelberg Retinal Tomograph II (HRT II, Heidelberg Engineering) is a non-invasive, confocal scanning laser imaging system that uses a red (670 nm) diode laser to perform a series of optical sections of the macula area covering a 15°x15° field of view, corresponding to approximately 4.5 x 4.5 mm on the retina. The reflected laser light intensity is processed assisting with a quantitative diagnosis of ME. If ME is present, the amount of scatter inside the swollen retina increases, reducing retinal reflectance.

A few studies have evaluated the HRT for detecting ME. Tong and co-workers have proposed a scoring system for macular image assessment using HRT in patients with diabetic maculopathy. Guan and co-workers found the HRT to have a sensitivity and specificity of 92% and 68% for detecting ME in the diabetic population when using clinical assessment as the gold standard. To the best of our knowledge, no studies have yet validate the used HRT for the detection of ME as an early sign of exudative disease in ARMD patients.

Purpose: The purpose of the study is to assessed the sensitivity, specificity, and repeatability, of HRT for the presence of ME in exudative ARMD Design: Prospective, observational study. Objectives: 1) Assessment of healthy volunteers to obtain baseline normal measurements of macular thickening. 2) Measurements in ARMD patient's referred to a retinal specialist clinic with the diagnosis of exudative form of ARMD Patients, Material, and Methods: 1) normal controls (N=20): baseline measurements centered at the fovea will be taken. Three consecutive measurements will be performed (within-session repeatability). 2) Patients: New patients referred by general ophthalmologists to the retina specialist for possible diagnosis of ARMD, exudative formed, will be included in the study. All patients will undergo a full ophthalmologic exam by the same retinal specialist who will determine the clinical presence of ME (gold standard) using fundus contact lens examination. In some cases, fluorescein angiograms will be use as an ancillary test. All patients will then be evaluated using HRT for the presence of ME using the macula edema module. The technician performing the test will be mask to the patients' clinical diagnosis. Three consecutive measurements will be performed in 4 quadrants (500-1000-1500 microns/ 4 quadrants) (color map and reflectivity) 3) Comparison will be made between the clinical diagnosis of ME (gold standard) and results obtained by the HRT. Features compared: 1) presence/absence of ME 2) spacial agreement between areas of elevated retina encountered by HRT Vs clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* New patients referred by general ophthalmologists to the retina specialist for possible diagnosis of ARMD, exudative formed, will be included in the study.

Exclusion Criteria:

* Significant media opacity
* Other causes of macular edema (ME) (diabetes, vascular occlusions)
* Diabetic patients with retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of screening test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mila Oh, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada